CLINICAL TRIAL: NCT00630565
Title: Autologous Peripheral Blood Stem Cell Transplant for Acute Non-Lymphocytic Leukemia (ANLL)
Brief Title: Stem Cell Transplant in Treating Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT2006-13; 0607M89052 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-03-06; First posted 2008-03-07 (Estimated); Results first posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(16;16)(p13;q22); childhood acute myeloid leukemia in remission
MeSH Terms: conditions — Leukemia; Congenital Abnormalities | interventions — sargramostim; Granulocyte Colony-Stimulating Factor; Busulfan; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; Etoposide; Bone Marrow Transplantation; Hematopoietic Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Bone Marrow Transplant (2-70 Years old) (Experimental): Patients over the age of two will receive a cytoreductive regimen of total-body irradiation and cyclophosphamide (TBI/CY) as well as sargramostim, dexamethasone, etoposide, transplantation (bone marrow transplantation/hematopoietic stem cell transplantation/peripheral blood stem cell transplantation).
  Interventions: Biological: sargramostim; Drug: cyclophosphamide; Drug: dexamethasone; Drug: etoposide; Procedure: bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation
- Bone Marrow Transplant (less and 2 years old) (Experimental): Patients under the age of two, and patients who cannot receive total body irradiation (TBI), will receive a cytoreductive regimen of Busulfan and cyclophosphamide (BU/CY) as per the Johns Hopkins University Hospital regimen as well as sargramostim, dexamethasone, etoposide, transplantation (bone marrow transplantation/hematopoietic stem cell transplantation/peripheral blood stem cell transplantation).
  Interventions: Biological: sargramostim; Drug: busulfan; Drug: cyclophosphamide; Drug: dexamethasone; Drug: etoposide; Procedure: hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: sargramostim — Given subcutaneously (SC) 10 μg/kg/day from day +3 until apheresis is completed
  Other Names: G-CSF
Drug: busulfan — 4 mg/kg po in 4 divided doses (.8 mg/kg/dose orally every 6 hours) on days -7 through -4.
  Other Names: Busulfex
  Arms: Bone Marrow Transplant (less and 2 years old)
Drug: cyclophosphamide — 4 gm/m^2 x 1 (day 0) and 60 mg/kg intravenous (IV) over 2 hours on days -3 and -2.
  Other Names: Cytoxan
Drug: dexamethasone — 20 mg/m^2 x 4 doses every 12 hours given intravenously (IV) push before cytoxan on day 0 and then every 12 hours
  Other Names: Decadron
Drug: etoposide — 300 mg/m^2/day x 2 days (day 0-1) over 3 hours intravenously (IV)
  Other Names: VP-16
Procedure: bone marrow transplantation — Day 0 infusion of bone marrow cells
  Other Names: ABMT
  Arms: Bone Marrow Transplant (2-70 Years old)
Procedure: hematopoietic stem cell transplantation — Stem cell infusion (>48 hours after the last dose of cyclophosphamide)
  Other Names: HSCT
  Arms: Bone Marrow Transplant (less and 2 years old)
Procedure: peripheral blood stem cell transplantation — Day 0 infusion of peripheral blood stem cells
  Other Names: PBSCT
  Arms: Bone Marrow Transplant (2-70 Years old)
Radiation: total-body irradiation — 165 cGy/dose given twice a day on days -7 through -4.
  Other Names: TBI
  Arms: Bone Marrow Transplant (2-70 Years old)

SUMMARY:
RATIONALE: Giving chemotherapy and colony-stimulating factors, such as G-CSF, may increase the number of stem cells in the blood. The stem cells are collected from the patient's blood and stored. Chemotherapy or radiation therapy is given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy.

PURPOSE: This clinical trial is studying how well an autologous stem cell transplant works in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess whether sufficient peripheral blood stem cells (PBSC) can be collected from patients with acute myeloid leukemia (AML) using cyclophosphamide, etoposide, and granulocyte-colony stimulating factor (G-CSF) mobilization.
* To assess the rate of myeloid, platelet, and erythroid recovery following autologous PBSC transplant.
* To assess the disease-free survival rate of patients with AML receiving PBSC auto grafts.

OUTLINE:

* Chemotherapy and filgrastim (G-CSF) priming for PBSC collection: Patients receive cyclophosphamide IV on day 0; etoposide IV over 3 hours on days 0 and 1; and oral dexamethasone twice daily on days 0 and 1. Patients also receive G-CSF subcutaneously (SC) beginning on day 3 and continuing until apheresis is complete. After blood counts recover, apheresis is performed in 4-6 daily planned collections until the minimum CD34+ cell dose of > 2.5 x 10^6 cells/kg is achieved. If the minimum CD34+ cell dose is not achieved after 6 apheresis collections, patients undergo bone marrow examination including a bone marrow biopsy and aspiration, at the termination of the PBSC collection to confirm remission. If remission is confirmed, and if peripheral counts and marrow cellularity are sufficient, the patient remains off G-CSF for 7 days and receives sargramostim (GM-CSF) for 5 days to increase the marrow cellularity, after which a bone marrow harvest is performed.
* Bone marrow harvest without prior PBSC collection: Children will undergo primed bone marrow harvest comprising GM-CSF IV or SC for 5 days prior to harvest to increase cellularity and then marrow is harvested. Marrow and blood specimens are also obtained with the initial bone marrow evaluation and at the time of harvest if a cytogenetic abnormality was previously described. Other patients who are unable to undergo PBSC collection may proceed with a bone harvest at the discretion of the protocol chairperson.
* Cytoreductive regimen:

  * Patients over 2 years old: Patients undergo total body irradiation (TBI) twice daily on days -7 to -4 (total of 8 fractions), cyclophosphamide IV over 2 hours on days -3 and -2, followed by a 1-day rest period on day -1.
  * Patients under 2 years old and patients who cannot undergo TBI: Patients receive busulfan IV or orally every 6 hours on days -7 to -4, cyclophosphamide IV over 2 hours on days -3 to -2, followed by a 1-day rest period on day -1.
* Stem cell transplantation: All patients undergo autologous PBSC and/or bone marrow infusion on day 0. Patients also receive G-CSF IV or SC beginning on day 1 and continuing until blood counts recover.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

Children under the age of two are eligible for this protocol, but will not receive total body irradiation. Instead, children under the age of two will receive Busulfan/Cyclophosphamide (Bu/Cy) conditioning as the preparative regimen in order to obviate deleterious effects of radiation at this age. Patients who cannot receive total body irradiation (TBI) (for example those with prior radiation therapy) will also receive the Bu/CY conditioning.

* Acute myeloid leukemia (AML)

  * All children and adults less than the age of 70 with AML who have achieved a first or second bone marrow remission are eligible for this protocol. Patients must undergo peripheral blood stem cell collection or marrow harvest while in remission and must not be expected to have better outcomes with allogeneic transplantation.
  * Patients with cytogenetic abnormalities suggesting an improved prognosis [t(8:21), t(15;17) and inv(16)] will be eligible for transplantation in first remission.
* Allogeneic transplant with an HLA-identical sibling will be recommended for patients <55 years. If the patient refuses allogeneic transplant, they may still be eligible for this protocol.

Exclusion Criteria:

* Patients can also be deemed not eligible for transplant because of specific organ toxicity. Specifically, patients with pre-existing compromise to the heart, lungs, kidney, CNS or liver may be excluded:

  * Eastern Cooperative Oncology Group (ECOG) Performance status: 0 or 1
  * Heart - The patient must be free of symptoms of uncontrolled cardiac disease, and must not have compromised cardiac function detected by ECHO or by gated cardiac blood flow scan (MUGA) LVEF >45%).
  * Kidney - The patient must have a corrected creatinine clearance >50% of normal.
  * Liver - The total serum bilirubin < 2.5 mg/dL; ALT <2 x upper limit of normal.
  * Lung - Patients must have no significant obstructive airways disease or resting hypoxemia (PO2 <80), and must have acceptable diffusion capacity (DLCO > 50% of predicted).
  * Central Nervous System (CNS): Patients must be free of active or ongoing ischemic or degenerative CNS disease and no active or resistant CNS leukemia.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-07-26 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Weisdorf, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone Marrow Transplant (2-70 Years Old) | Bone Marrow Transplant (Less and 2 Years Old)
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants enrolled under the age of 2 years old.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Marrow Transplant (2-70 Years Old) | Bone Marrow Transplant (Less and 2 Years Old) | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 0 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 6 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 0 | 8
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 0 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Engraftment
Description: Percentage of Participants with Engraftment measured by myeloid, platelet, and erythroid recovery
Time Frame: 30 Days Post Transplant
Measure: Number (95% Confidence Interval); unit: Participants of participants
Arm/Group | Bone Marrow Transplant (2-70 Years Old)
Number analyzed (Participants) | 12
Participants of participants | 100 [76 to 100]

2. Secondary Outcome: Percentage of Participants With Disease Response
Description: Disease evaluation will be completed approximately 100 days after stem cell infusion and every 6 months, 1 year, and until 2 years after infusion.
Time Frame: 2 years Post Transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bone Marrow Transplant (2-70 Years Old)
Number analyzed (Participants) | 12
Percentage of participants | 83 [46 to 95]

3. Secondary Outcome: Treatment Failure
Description: Percentage of participants experiencing treatment failure.
Time Frame: 2 years Post Transplant
Measure: Number; unit: Percentage of participants
Arm/Group | Bone Marrow Transplant (2-70 Years Old)
Number analyzed (Participants) | 12
Percentage of participants | 25

4. Secondary Outcome: Percent of Patients With Various Late Effects
Description: Description: (e.g., thyroid function abnormalities - T4, TSH, gonadal abnormalities, cataracts, pulmonary dysfunctions, growth and development abnormalities, and second malignant neoplasms)
Time Frame: 2 years Post Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Transplant (2-70 Years Old)
Number analyzed (Participants) | 12
Participants | 0

5. Secondary Outcome: Disease-free Survival
Description: Disease-free survival 2 years Post Transplant
Time Frame: 2 years Post Transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants with DFS
Arm/Group | Bone Marrow Transplant (2-70 Years Old)
Number analyzed (Participants) | 12
Percentage of participants with DFS | 73 [38 to 91]

6. Secondary Outcome: Percentage of Patients With Adequate Cells Collected
Description: The proportion of primed patients with adequate number of cells collected will be calculated.
Time Frame: Pre-Transplant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bone Marrow Transplant (2-70 Years Old)
Number analyzed (Participants) | 12
Percentage of participants | 75 [47 to 91]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Bone Marrow Transplant (2-70 Years Old)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Transplant (2-70 Years Old) (N=12)
Relapse (Blood and lymphatic system disorders) | 1 (1) — Relapse of acute promyelocytic leukaemia (APL)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT00630565/Prot_000.pdf
  • Informed Consent Form (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT00630565/ICF_001.pdf